CLINICAL TRIAL: NCT06323291
Title: Cancer Coaching and Remote Education for Self-Empowerment (CARES) Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Canopy Cancer Collective (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MCC-23077
Record Dates: First submitted 2024-03-14; First posted 2024-03-21 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Pancreatic Cancer
Keywords: Pancreas; Pancreatic Cancer; Caregiver
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Health Coaching for Pancreatic Cancer Patients (Other): Initial in-person and/or virtual supportive care, social work, and dietitian consultation within 4 weeks of diagnosis and/or 3 weeks of study enrollment.
  Interventions: Behavioral: Coaching Sessions
- Digital Health Coaching for Caregivers (Other): Initial in-person and/or virtual supportive care, social work, and dietitian consultation within 4 weeks of diagnosis and/or 3 weeks of study enrollment.
  Interventions: Behavioral: Coaching Sessions

INTERVENTIONS:
Behavioral: Coaching Sessions — Enrolled participants will set up an account through a secure and encrypted web portal managed by Osara Health.
  Coaches will follow-up with their designated patients and/or caregivers to schedule individual coaching sessions via phone, text, or email depending on the participant's communication preference. Participants will have an initial coaching consultation by phone to go over the purpose and structure of coaching sessions.
  Participants will then have an additional 3-4 coaching sessions (depending on time availability and need) to discuss symptom management, nutrition and exercise, sleep, and mindfulness.
  Participants will receive content for each of the modules via email.

SUMMARY:
This Pilot Study will evaluate a 12-week pilot program that offers digital health coaching for individuals with pancreatic cancer and their caregivers.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Participant must have a pancreatic cancer diagnosis or be a caregiver such as a friend or spouse.
* Participant must be planning to receive treatment and/or care management at Moffitt Cancer Center.
* Participant must be able to speak and read English.
* Participant must be able to provide informed consent.

Exclusion Criteria:

* Documented or observable psychiatric or neurological disorder that would interfere with study participation such as severe dementia
* Any participant that does not meet all inclusion criteria will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-05-26 (Actual); Study Completion 2025-05-26 (Actual)

PRIMARY OUTCOMES:
Recruitment Rate | Up to 12 Months
  Measured by ≥ 50% of eligible participants recruited.
Participant Acceptance of the Digital Health Coaching Program | Up to 12 Weeks
  Measured by ≥ 70% of participant rating of the intervention as satisfactory. 4 item scale (score range 0-20) will be utilized.
Participant Ease of Usability of the Digital Health Coaching Program | Up to 12 Weeks
  Measured by ≥ 70% of participant rating the mobile application as easy-to-use for scheduling coaching visits.
  4 item scale (score range 0-20) will be utilized.
Feasibility of Utilizing the Digital Health Coaching Program | Up to 12 Weeks
  Measured by ≥ 70% of participant rating of being likely to utilize the intervention.
  4 item scale (score range 0-20) will be utilized.

CONTACTS AND LOCATIONS:
Overall Officials: Amir Alishahi Tabriz, MD, PhD, Principal Investigator — Moffitt Cancer Center; Pamela Hodul, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials Website — http://www.moffitt.org/clinical-trials-research/clinical-trials/